CLINICAL TRIAL: NCT06640478
Title: NUTRI-Beta Study: A Pilot Clinical Trial for Children With New Diagnosis of Stage 3 Type 1 Diabetes
Brief Title: A 12-week Pilot Nutrition Intervention for Children With New Diagnosis of Stage 3 Type 1 Diabetes (T1D)
Acronym: NUTRI-Beta
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Lina Huerta-Saenz, Assistant Professor Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00020631
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: T1D; Healthy foods; Children; Youth; Nutrition Counseling; Diabetes mellitus type 1; Nutrition; Honeymoon phase; partial remission of diabetes; new diagnosis of type 1 diabetes; healthy eating; Nutrition Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Sub-investigators, research assistants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTRI-Beta Intervention Group (Active Comparator): We will provide healthy foods (NUTRI-Beta Food bag) to the intervention group weekly for 12 weeks, in addition to an intensive nutrition counseling program (NUTRI-Beta Counseling) and close 24-hour continuous glucose monitoring. The healthy foods bag will contain a combination of 6 types of foods including:
  1. seasonal fruits (containing high amounts of vitamin C and E)
  2. legumes,
  3. nuts,
  4. yogurt, and
  5. seasonal vegetables (carotenoids, tomatoes, broccoli, celery, etc.).
  6. seafood or seafood-related products
  The portions of each food group component of the NUTRI-Beta basket will follow the current USDA dietary guidelines according to the age of the participant: a) Intervention group will receive NUTRI-Beta foods bag + intensive nutrition counseling (NUTRI-Beta dietary counseling) + standard insulin treatment (either insulin injections or insulin pump per patient preference) and T1D technology use
  Interventions: Other: NUTRI-Beta Counseling; Dietary Supplement: Free weekly produce foods
- Standard of care nutrition counseling (MyHealthy plate model and ADA clinical guidelines) (Other): STANDARD OF CARE NUTRITION COUNSELING:
  1. A 12-week distribution of weekly grocery store gift cards of similar monetary value of the NUTRI-Beta food bag in addition to
  2. MyPlate USDA model with similar frequency of nutrition counseling visits but following the American Dietary Association (ADA) Guidelines, and
  3. Standard insulin treatment (either insulin injections or insulin pump per patient preference) and 24-hour continuous glucose monitor
  Interventions: Dietary Supplement: Standard dietary counseling

INTERVENTIONS:
Other: NUTRI-Beta Counseling — Dietary Counseling focused on anti-inflammatory foods
  Other Names: NUTRI-Beta Intervention
  Arms: NUTRI-Beta Intervention Group
Dietary Supplement: Standard dietary counseling — Standard of Care therapy: Nutrition counseling per the ADA clinical guidelines and USDA MyPlate model
  Other Names: Standard
  Arms: Standard of care nutrition counseling (MyHealthy plate model and ADA clinical guidelines)
Dietary Supplement: Free weekly produce foods — Free weekly produce
  Arms: NUTRI-Beta Intervention Group

SUMMARY:
The purpose of this research study is to investigate the effects of a combination of weekly distribution of healthy foods and intensive nutrition counseling as complementary therapies to the standard insulin therapy in children with new diagnosis of stage 3 type 1 diabetes (T1D). Feasibility, acceptability, and fidelity of this intervention will be measured. We will also explore the likelihood of prolonging the honeymoon phase of T1D in the intervention study group. Comparisons will be made between this combined nutrition intervention and free healthy foods vs. current standard nutrition counseling. Both study groups will receive standard of care treatment for T1D (insulin therapy).

The results of this study could inform future research that will ultimately lead to design of a larger clinical trial testing implementation of novel medical nutrition therapies for children newly diagnosed with stage 3 of T1D, and may lead to prolongation of the honeymoon phase. The overall goal is to promote the beta cell function survival and to reduce the progression to stage 4 of T1D.

Condition or Disease:

* Type 1 Diabetes Mellitus
* New Diagnosis of Stage 3 Type 1 Diabetes ≤ 60days

Intervention/Treatment:

- Weekly Free Healthy Foods + Intensive Nutrition Counseling for 12 weeks

DETAILED DESCRIPTION:
The proposed study is a 12-week pilot, single-blinded, randomized, controlled clinical trial in prepubertal children (6-17 years old) newly diagnosed with stage 3 of type 1 diabetes (T1D) within 60 days. The total duration of the study is 24 weeks, but the nutrition intervention is only delivered during 12 weeks with a 24-week follow up visit. We expect to enroll a total of 12-40 children (6-20 per study group).

We will be investigating the potential role of a frequent personalized nutrition counseling intervention (7 sessions in a hybrid model) in addition to weekly distribution of selected healthy foods. We expect the diet quality of the youth receiving the intervention (you) will improve during and after the study intervention.

There will be two study groups: intervention and control group.

The intervention group will receive a food bag containing specific healthy foods with high anti-inflammatory properties weekly for 12 weeks, in addition to seven nutrition counseling sessions. The provided foods are a combination of 6 types of foods including: a) seasonal fruits (containing high amounts of vitamin C and vitamin E), b) legumes, c) nuts, d) yogurt, e) vegetables and f) seafood. The portions of each food group component of the "healthy foods bag" will follow the current USDA dietary guidelines according to the age of the study participant. [1] By contrast, the control group will receive weekly grocery store gift cards of similar monetary value of the "healthy food bag" in addition to seven nutrition counseling sessions based on the standard MyHealthy plate model.

In regards to the nutrition counseling sessions, this counseling will be provided as a hybrid model with a combination of 4 in-person nutrition counseling sessions and 3 virtual dietary counseling sessions provided by a registered dietitian. In summary:

1. Intervention group will receive NUTRI-Beta foods basket + nutrition counseling (NUTRI-Beta dietary counseling) + standard insulin treatment (either insulin injections or insulin pump per patient preference)+ standard of care insulin therapy and use of a 24-hour continuous glucose monitor, and
2. Control group will receive the standard nutrition counseling per the American Dietary Association (ADA) Guidelines [2] + weekly grocery store gift cards + standard of care insulin therapy and use of a 24-hour continuous glucose monitor.

The NUTRI-Beta clinical trial study visits will include a total of 10 visits during the 24 weeks of the study: Screening visit (V0), baseline visit (enrolment visit= V1), nutrition counseling visit 2 (week 2 post enrollment), nutrition counseling visit 3 (V3-virtual, week 3), nutrition counseling visit 4 (V4-in person, week 4), nutrition counseling visit 5 (V5-virtual, week 6), nutrition counseling visit 6 (V6-in person, week 8), nutrition counseling visit 7 (V7-virtual, week 10), visit 8 ( 12 weeks after enrollment- end of nutrition intervention), and visit 9 (24 weeks after enrollment).

We expect that this nutrition intervention (NUTRI-Beta) will be acceptable to children with new diagnosis of clinical diabetes (stage 3 of T1D) and will improve their diet intake and quality, their nutrition status and may increase their likelihood of residual beta-cell function in the treatment group. Evaluation of the partial remission of T1D will be completed through the determination of the insulin dose-adjusted A1C (IDAA1C) and residual beta cell function through the measurement of peak C-peptide levels during a 2-hour mixed-meal tolerance test (MMTT) after 12 and 24 weeks of the nutrition intervention.

The treatment group is expected to have higher rates of partial remission of T1D measured by the IDAA1C, better diet quality, better glycemic metrics and reduced needs of total daily dose of insulin (TDD) (unit/kg/day).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give assent and to have a parent or legal guardian to provide informed consent
2. Less or equal than 60 days from T1D diagnosis based on American Diabetes Association criteria, and metabolically stable per study physician assessment
3. Boys and girls (Any Tanner stage), 6-17 years of age, at time of enrollment visit
4. Evidence of at least one positive T1D autoantibody (excluding insulin antibodies in those who have received ≥ 2 weeks of exogenous insulin therapy) either through clinically obtained labs at time of diagnosis or as obtained at the screening visit
5. Children with new diagnosis of T1D need to be established patients from Penn State Health- Pediatric diabetes clinic at the time of the enrollment visit
6. Capability to eat different types of food by mouth
7. Daily use of a 24-hour continuous glucose monitor by the time of the enrollment visit
8. Willing and being able to give assent and have a parent or legal guardian provide informed consent

Exclusion Criteria:

1. Children with new diagnosis of T1D who are not metabolically stable (E.g. acute dehydration, severe hyperglycemia with moderate/large ketones at the time of the enrollment visit)
2. Concurrent or recent (within the past 30 days of screening) use of non-insulin therapies to control hyperglycemia including immunosuppressive therapies
3. Chronic inflammatory or autoimmune diseases with exception of stable autoimmune thyroid disease
4. Children requiring enteral feeds or parenteral nutrition support
5. Diagnosis of celiac disease or being actively evaluated for possible celiac disease, inflammatory bowel disease or any underlying illness cause acute or chronic intestinal malabsorption.
6. Use of glucocorticoids or other immunosuppressive agents within 30 days of T1D diagnosis
7. Use of medications known to influence glucose intolerance within 30 days of T1D diagnosis
8. Food allergies (nuts, soy, seafood, milk-protein, or as deemed by the principal investigator) that are a barrier for consumption of a balanced diet that meets nutrient requirements
9. Prior diagnosis or positive screening of food sensory disorders
10. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation to the study results

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 6 months
  Number of subjects screened over the course of the study
Enrollment rates | 6 months
  Number of subjects participating over the course of the study
Amount of time required to recruit the target sample (approx. 12- 20 people) | 6 months
  Number of months necessary to meet recruitment goals
Number of subjects required to be screened to meet required sample size (approx. 12- 20 people) | 6 months
  Number of subjects screened to meet enrollment goals
Number of participants who completed the 12-week intervention | 12 weeks
  Number of subjects completing the intervention
Average number of provided foods consumed during the day over the course of the intervention | 12 weeks
  Average number of provided foods consumed during the day over the course of the intervention
Number of participants who completed the Mixed-meal tolerance test at the enrollment visit | Baseline
  Number of subjects completing the MMTT at baseline
Number of participants who completed the Mixed-meal tolerance test at the 12-week visit | 12 weeks
  Number of subjects completing the MMTT at 12 week visit
Number of participants who completed the Mixed-meal tolerance test at the 24-week visit | 24 weeks
  Number of subjects completing the MMTT at 24 week visit

SECONDARY OUTCOMES:
Healthy Eating Index (HEI) change from baseline to the 12-week visit | 12 weeks
  HEI ranges from 0-100, with an ideal score being 100.
Healthy Eating Index (HEI) change from baseline to the 24-week visit. | 24 weeks
  HEI ranges from 0-100, with an ideal score being 100.
Weight changes from baseline visit to the 12-week visit | 12weeks
  Change in subject weight
Weight changes from baseline visit to the 24-week visit | 24 weeks
  Change in subject weight
Weight Z-score changes from baseline visit to the 12 week visit | 12 weeks
  Change in subject weight z-score
Weight Z-score changes from baseline visit to the 24 week visit | 24 weeks
  Change in subject weight z-score
Height changes from baseline to the 12 week visit | 12 weeks
  Change in subject height
Height changes from baseline to the 24 week visit | 24 weeks
  Change in subject height
Height Z-score changes from baseline to the 12 week visit | 12 weeks
  Change in subject height z score
Height Z-score changes from baseline to the 24 week visit | 24 weeks
  Change in subject height z score
Body Mass Index (BMI) changes from baseline to the 12 week visit | 12 weeks
  Change in subject BMI
Body Mass Index (BMI) changes from baseline to the 24 week visit | 24 weeks
  Change in subject BMI
BMI Z-score changes from baseline to 12 weeks | 12 weeks
  Change in subject BMI z-score
BMI Z-score changes from baseline to 24 weeks | 24 weeks
  Change in subject BMI z-score
Height velocity changes from baseline visit to the 12-week visit | 12 weeks
  Change in subject height velocity
Height velocity changes from baseline visit to the 24-week visit | 24 weeks
  Change in subject height velocity
Percentage of time in range (TIR) glucose levels from baseline to 3 month intervention visit | 3 months
  Change in percentage of TIR glucose levels from baseline to 3 month intervention visit
Percentage of time in range (TIR) glucose levels from baseline to 6-month post intervention visit | 24 weeks
  Change in percentage of TIR glucose levels from baseline to 24-week visit
Percentage of time above range (TAR) glucose levels from baselines to 3 month intervention visit | 3 months
  Change in percentage of TAR glucose levels from baseline to 3 month intervention visit
Percentage of time above range (TAR) glucose levels from baseline to the 6 -month post intervention visit | 6 months
  Change in percentage of TAR glucose levels from baseline to 6 month post intervention visit
Percentage of time below range (TBR) glucose levels from baselines to 3 month intervention visit | 3 months
  Change in percentage of TBR glucose levels from baseline to 3 month intervention visit
Percentage of time below range (TBR) glucose levels from baselines to 6 month post intervention visit | 6 months
  Change in percentage of TBR glucose levels from baseline to 6 month post intervention visit
Percentage of mean glucose level from baseline to 12-week visit | 12 weeks
  Change in percentage of mean blood glucose level from baseline to 12-week visit
Percentage of average glucose levels from baseline to 6 month post intervention visit | 6 months
  Change in percentage of average glucose levels from baseline to 6 month post intervention visit
Percentage of standard deviation of glucose levels from baseline to 3 month intervention visit | 3 months
  Change in percentage of standard deviation glucose levels from baseline to 3 month intervention visit
Percentage of standard deviation of glucose levels from baseline to 6 month post intervention visit | 6 months
  Change in percentage of standard deviation of glucose levels from baseline to 6 month post intervention visit
Percentage of coefficient of variation (CV) of glucose levels from baseline to 3 month intervention visit | 3 months
  Change in percentage of CV of glucose levels from baseline to 3 month intervention visit
Percentage of coefficient of variation (CV) of glucose levels from baseline to 6 month post intervention visit | 6 months
  Change in percentage of CV of glucose levels from baseline to 6 month post intervention visit
Percentage of glucose management index (GMI) of glucose levels from baseline to 3 month intervention visit | 3 months
  Change in percentage of GMI of glucose levels from baseline to 3 month intervention visit
Percentage of glucose management index (GMI) of glucose levels from baseline to 6 month post intervention visit | 6 months
  Change in percentage of GMI of glucose levels from baseline to 6 month post intervention visit
Percentage of hemoglobin A1C (HbA1C) of glucose levels from baseline to 3-month intervention visit | 3 months
  Change in percentage of HbA1C glucose levels from baseline to 3-month intervention visit
Percentage of hemoglobin A1C (HbA1C) of glucose levels from baseline to 6 month post intervention visit | 6 months
  Change in percentage of HbA1C glucose levels from baseline to 6 month post intervention visit
Dietary intake changes on daily total K- calories from baseline visit to 12 week visit | 12 weeks
  Change in dietary intake on daily total K-calories will be obtained through the use of the ASA24 dietary online tool, measuring daily total K-calories.
Dietary intake changes on daily total K- calories from baseline visit to 24 week visit | 24 weeks
  Change in dietary intake on daily total K-calories will be obtained through the use of the ASA24 dietary online tool, measuring daily total K-calories.
Macronutrient intake composition from baseline to 12 week visit | 12 weeks
  Change in macronutrient intake composition will be obtained through the use of the ASA24 dietary online tool, measuring daily percentage of macronutrients (carbohydrates, proteins, and fats)
Macronutrient intake composition from baseline to 24 week visit | 24 weeks
  Change in macronutrient intake composition will be obtained through the use of the ASA24 dietary online tool, measuring daily percentage of macronutrients (carbohydrates, proteins, and fats)
Micronutrient intake composition from baseline to 12 week visit | 12 weeks
  Change in micronutrient intake composition will be obtained through the use of the ASA24 dietary online tool, measuring daily percentage of micronutrients
Micronutrient intake composition from baseline to 24 week visit | 24 weeks
  Change in micronutrient intake composition will be obtained through the use of the ASA24 dietary online tool, measuring daily percentage of micronutrients
Changes in the baseline levels of carotenoids, vitamin C and vitamin E | 12 weeks
  Changes in levels of carotenoids, vitamin C and vitamin E from baseline to 12-week visit
Changes in the baseline levels of carotenoids, vitamin C and vitamin E | 24 weeks
  Changes in levels of carotenoids, vitamin C and vitamin E from baseline visit to 24-week visit
Changes on the levels of 25-hydroxy vitamin D | 12 weeks
  Changes on the baseline level of 25-hydroxy vitamin D level to the 12-week visit
Changes on the levels of 25-hydroxy vitamin D | 24 weeks
  Changes on the baseline level of 25-hydroxy vitamin D level to 24-week visit
Omega 3 index (O3i) levels changes during the clinical trial | 12 weeks
  Changes of baseline levels of Omega 3 index (O3i) to 12-week visit
Omega 3 index levels during clinical trial | 24 weeks
  Changes of Omega 3 index level from baseline visit to the 24-week study visit
Middle Upper Arm Circumference (MUAC) changes | 12 weeks
  Middle Upper Arm Circumference (MUAC) changes From enrollment visit to 12-week visit (end of nutrition intervention)
Middle Upper Arm Circumference (MUAC) | 24 weeks
  Middle Upper Arm Circumference (MUAC) changes from enrollment visit to 24-week visit (end of the study)

OTHER OUTCOMES:
Area under the curve and peak C-peptide level determined by MMTT (Mixed Meal Tolerance Test) | 2 hours
  Peak c-peptide levels from baseline over the course of 2 hours
Change in the total daily dose of exogenous insulin (TDD) as units/kg/day from baseline to the 12-week visit | 12 weeks
  Change in TDD of insulin
Change in the total daily dose of exogenous insulin (TDD) as units/kg/day from baseline to the 24-week visit. | 24 weeks
  Change in TDD of insulin
Change in the IDAA1C from enrollment (baseline) visit to the 12-week study visit | 12 weeks
  Change in the IDAA1C
Change on the IDAA1C from enrollment (baseline) visit to the 24-week study visit | 24 weeks
  Change in the IDAA1C

CONTACTS AND LOCATIONS:
Overall Officials: Lina Huerta Saenz, MD, FAAP, Principal Investigator — Pediatric Endocrinologist, Assistant Professor of Pediatrics, Penn State Health Milton Hershey Medical Center, Penn State College of Medicine
Locations (2):
- United States (2):
  - Penn State Health Children's, Hershey, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania